CLINICAL TRIAL: NCT05402943
Title: The Effect of Nursing Care Program Developed Based on Health Promotion Model on the Healthy Lifestyle Behaviors and Quality of Life of Women With Endometriosis.
Brief Title: The Effect of Nursing Care Program on Women With Endometriosis
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ayse Gul BURSA, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: IST.UNI.CERRAH.DEPT.OF NURSING
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Endometriosis; Quality of Life; Healthy Life Style
Keywords: Endometriosis, Health Promotion Model, Nursing Care
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: The group which interventions applied during study.
  Interventions: Behavioral: Nursing Care Program for Endometriosis; Behavioral: EHP-5 Endometriosis Health Promotion Model.; Behavioral: Healthy Life Style Behaviours Scale II.; Behavioral: The Satisfaction Questionnaire for Nursing Care Program for women with Endometriosis.
- Control Group: None intervention applied.
  Interventions: Behavioral: EHP-5 Endometriosis Health Promotion Model.; Behavioral: Healthy Life Style Behaviours Scale II.

INTERVENTIONS:
Behavioral: Nursing Care Program for Endometriosis — Nursing Care Program for Endometriosis, developed in line with Health Promotion Model
  Groups: Intervention Group
Behavioral: EHP-5 Endometriosis Health Promotion Model. — EHP-5 Endometriosis Health Promotion Model. A questionnaire used to measure the quality of life of women with endometriosis
Behavioral: Healthy Life Style Behaviours Scale II. — A questionnaire used to measure the Healthy Life Style Behaviours.
Behavioral: The Satisfaction Questionnaire for Nursing Care Program for women with Endometriosis. — A questionnaire used to measure the satisfaction levels of women with endometriosis who applied the Nursing Care Program for women with endometriosis.
  Groups: Intervention Group

SUMMARY:
This study was carried out to determine the effect of the endometriosis nursing care program (ENCP) given to women with endometriosis in line with the Health Promotion Model, on the quality of life and healthy lifestyle behaviors of women.

DETAILED DESCRIPTION:
This experimental study, which was conducted in a single-blind, with control group, prospective, randomized type in the first test-post-test order, was carried out in the endometriosis polyclinic of Istanbul Zeynep Kamil Gynecology and Pediatrics Training and Research Hospital.

In the preliminary evaluation, 46 women with Endometriosis Health Profile Questionnaire-5 (EHP-5) scores of 22 and above (50 and above in the 100 system) constituted the sample of the study, including 23 intervention and 23 control groups. While the Nursing Care Program for Women with Endometriosis (NCPE) was applied to the intervention group, only routine care was applied to the control group. Introductory Information Form, EHP-5, Healthy Lifestyle Behaviors Scale II (HLBSII), and Satisfaction Questionnaire for NCPE were used as data collection forms in the study.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with endometriosis,
* Being in the reproductive period,
* No communication barrier,
* Not having been diagnosed with a psychiatric illness,

Exclusion Criteria:

* Getting pregnant during the study,
* It was determined as wanting to leave the study,

Ages: 25 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women diagnosed with endometriosis who applied to the outpatient clinic.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
The quality of life assessed by the EHP-5 | May 2021-June 2022
  The quality of life of women with endometriosis is assessed by Endometriosis Health Profile Questionnaire-5 .
Healthy lifestyle behaviours assessed by the HLBS II. | May 2021-June 2022
  The healthy lifestyle behaviours of women with endometriosis is assessed by Healthy Lifestyle Behaviors Scale II (HLBSII).

SECONDARY OUTCOMES:
Satisfaction level of women assessed by questionnaire developed in line with the literature. | May 2021-June 2022
  The Satisfaction levels measured with a questionnaire developed in line with the literature, of the women in the intervention group who were applied Nursing Care Program for Women with Endometriosis (NCPE), developed by researcher in line with the Health Promotion Model.

CONTACTS AND LOCATIONS:
Overall Officials: Nevin SAHIN, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul Zeynep Kamil Women and Children Disease Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones G, Kennedy S, Barnard A, Wong J, Jenkinson C. Development of an endometriosis quality-of-life instrument: The Endometriosis Health Profile-30. Obstet Gynecol. 2001 Aug;98(2):258-64. doi: 10.1016/s0029-7844(01)01433-8. PMID 11506842
- [Background] Jones G, Jenkinson C, Kennedy S. Development of the Short Form Endometriosis Health Profile Questionnaire: the EHP-5. Qual Life Res. 2004 Apr;13(3):695-704. doi: 10.1023/B:QURE.0000021321.48041.0e. PMID 15130031
- [Background] Walker, S. N., & Hill-Polerecky, D. M. (1996). Psychometric evaluation of the health- promoting lifestyle profile II. Unpublished manuscript, University of Nebraska Medical Center, 120-26..
- [Background] Selcuk S, Sahin S, Demirci O, Aksoy B, Eroglu M, Ay P, Cam C. Translation and validation of the Endometriosis Health Profile (EHP-5) in patients with laparoscopically diagnosed endometriosis. Eur J Obstet Gynecol Reprod Biol. 2015 Feb;185:41-4. doi: 10.1016/j.ejogrb.2014.11.039. Epub 2014 Dec 4. PMID 25522117
- [Background] Bahar, Z., Beşer, A., Gördes, N., Ersin, F., & Kıssal, A. (2008). Sağlıklı Yaşam Biçimi Davranışları Ölçeği II'nin geçerlik ve güvenirlik çalışması. C.Ü. Hemşirelik Yüksekokulu Dergisi, 12(1)
- [Background] D'Alterio, M. N., Saponara, S., Agus, M., Laganà, A. S., Noventa, M., Loi, E. S., Feki, A., & Angioni, S., 2021, Medical and surgical interventions to improve the quality of life for endometriosis patients: A systematic review, Gynecological Surgery 18(1), 1-14. https://doi.org/10.1186/s10397-021-01096-5.
- [Background] De Graaff AA, D'Hooghe TM, Dunselman GA, Dirksen CD, Hummelshoj L; WERF EndoCost Consortium; Simoens S. The significant effect of endometriosis on physical, mental and social wellbeing: results from an international cross-sectional survey. Hum Reprod. 2013 Oct;28(10):2677-85. doi: 10.1093/humrep/det284. Epub 2013 Jul 11. PMID 23847114
- [Background] Fedele, F., 2021, An Overview on the Psychological Impact of Endometriosis on Adolescent Girls' Life, Women's Health Bulletin. https://doi.org/10.30476/whb.2021.91557.1128.
- [Background] Fourquet J, Baez L, Figueroa M, Iriarte RI, Flores I. Quantification of the impact of endometriosis symptoms on health-related quality of life and work productivity. Fertil Steril. 2011 Jul;96(1):107-12. doi: 10.1016/j.fertnstert.2011.04.095. Epub 2011 May 31. PMID 21621771